CLINICAL TRIAL: NCT03789968
Title: The Incidence and Severity of Drug Interactions Before and After Switching Antiretroviral Therapy to Bictegravir/Emtricitabine/Tenofovir Alafenamide in Treatment Experienced Patients
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: University of Maryland, College Park (Other); Indiana University Health (Other); The Brooklyn Hospital Center (Other); University of Illinois at Chicago (Other); Nova Southeastern University (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Jason Schafer, Associate Professor, Department of Pharmacy, Thomas Jefferson University
Other Study IDs: 18G.786
Record Dates: First submitted 2018-12-26; First posted 2018-12-31 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: bictegravir/emtricitabine/tenofovir alafenamide — Treatment experienced patients with HIV infection that switched to a bictegravir/emtricitabine/tenofovir alafenamide-based ART regimen

SUMMARY:
This study will assess changes in the incidence and severity of drug interactions before and after switching antiretroviral therapy to bictegravir/emtricitabine/tenofovir alafenamide-based regimens in treatment experienced patients living with HIV infection.

DETAILED DESCRIPTION:
Simple, safe and effective antiretroviral therapy (ART) can provide optimal treatment outcomes for people living with HIV infection (PLWH) [1]. Increasingly complex and poorly tolerated regimens, on the other hand often limit ART adherence, while drug-drug interactions (DDIs) and safety concerns with individual ART agents can limit treatment selection [2-4]. Fortunately, recent advances in ART have included the emergence of several highly effective, safe and well tolerated regimens with limited DDIs. In clinical trials, integrase strand transfer inhibitors (INSTIs) such as raltegravir, elvitegravir, dolutegravir and bictegravir are consistently as effective or more effective than comparator agents and often superior in terms of tolerability [5-10]. Due to their efficacy, safety, and tolerability, INSTI-based regimens are now routinely used in treatment naïve patients and emerging data suggests that several may be used to simplify therapy for selected patients with treatment experience [11, 12].

Among the INSTIs, bictegravir is the newest agent in the class [13]. Similar to dolutegravir and raltegravir and in contrast to elvitegravir, it has few significant drug-drug interactions. Unlike dolutegravir and raltegravir, bictegravir is available as part of a single-tablet, once-daily regimen that includes tenofovir alafenamide and emtricitabine (BIC/TAF/FTC). Raltegravir is not available within a single tablet regimen, while dolutegravir is available as part of a single-tablet regimen, but it includes abacavir, which has been linked to an increased cardiovascular disease risk. As a result, BIC/TAF/FTC is currently among the most effective, safe, well-tolerated treatment options with limited drug-drug interactions.

With several new treatment options available, particularly in the INSTI class, current guidelines advocate switching ART when possible in virologically suppressed, ART experienced patients [1]. Switching ART can simplify treatment, improve tolerability, eliminate toxicity, and mitigate drug-drug interactions. When switching ART for any reason, it is critical to review a patient's full HIV treatment history, including virologic responses, past ART-associated toxicities, and cumulative resistance before selecting a new regimen [1].

Drug-drug interaction assessments with a patient's concomitant medications should also be performed prior to switching ART. More than 70% of the HIV population will be above the age of 50 by the year 2020 and many are receiving 5 or more medications for common chronic conditions in addition to being ART experienced [14, 15]. Cardiovascular disease, hepatic and renal disease, osteoporosis, insulin resistance, metabolic disorders, and cancers are among the conditions that can occur more commonly in PLWH and at times earlier in life in comparison to their HIV negative counterparts [16]. Drug-drug interactions between medications needed to treat or prevent these comorbid conditions can often interact with ART. Switching ART, in many circumstances can reduce the number drug interactions with medications for comorbid conditions. Conversely, switching can also lead to new interactions requiring intervention to avoid toxicities or prevent ineffective treatment.

Multiple studies have confirmed that switching HIV treatment can improve patient adherence and quality of life [17]. Several studies have also confirmed that clinically significant drug-drug interactions are common in patients living with HIV, but none have assessed changes in the incidence and severity of drug-drug interactions in the setting of ART switches [18-20]. The primary objective of this study is to assess changes in the incidence and severity of drug interactions before and after switching ART to BIC/TAF/FTC -based regimens in treatment experienced patients.

Null Hypothesis:

There is no difference in the incidence and severity of drug-drug interactions between ART and concomitant medications before and after switching to a BIC/TAF/FTC-based ART regimen in treatment experienced patients.

Alternative Hypothesis:

The incidence and severity of drug-drug interactions between ART and concomitant medications is reduced after switching to a BIC/TAF/FTC-based ART regimen in treatment experienced patients.

Data Collection Subjects from the Jefferson Infectious Diseases Associates outpatient HIV Clinic will be evaluated for study inclusion. Co-investigators at six partner institutions will also evaluate patients at their HIV clinics for study inclusion. The following information will be collected for patients meeting the study criteria: age, gender, race, duration of HIV infection, duration of ART treatment, number of previous ART regimens, CD4+ cell count and HIV RNA directly prior to switching to a BIC/TAF/FTC-based ART regimen, and the reason for switching ART to a BIC/TAF/FTC-based regimen. Additionally, all concomitant medication names at the time of the ART switch will be collected.

Scoring System To assess the combined incidence and severity of drug interactions with concomitant medications (CM) prior to and following each patient's ART switch, a DDI incidence and severity score was developed. The score is based upon results obtained when entering medications into the University of Liverpool's HIV Drug Interaction Checker (ULHDIC) database [21]. Each ART-CM pair is given one of the following scores: "do not co-administer" is assigned a score of 2, "potential interaction" a score of 1, and "potential weak interaction" or "no interaction" a score of 0. For those interactions that have "no clear data," or for those medications that are not listed in the drug database, the Department of Health and Human Services HIV treatment guidelines will be consulted along with the FDA product labeling.

Score Validation A separate analysis (data not provided here) was completed by study investigators to validate the use of the ULDIC severity ranking. The medication profiles of a random, representative sample of the study's population were selected for analysis. Drug interaction scores using the aforementioned ULHDIC were compared with drug interaction scores determined manually using the Department of Health and Human Services HIV treatment guidelines and FDA product labeling. No statistical difference in drug interaction scores between methods was observed.

Primary Endpoint The primary endpoint of the study will be to measure the change in mean total drug interaction scores pre and post ART switch to a BIC/TAF/FTC-based ART regimen. The total drug interaction scores for each patient pre- and post-switch will be calculated. The average pre-switch and post-switch scores will then be determined and analyzed for statistical differences using a two-sided paired t-test (normal distribution) with an alpha level of 0.05 or a Wilcoxon Ranked Sum test (non-normal distribution).

Secondary Endpoints The secondary endpoint of the study will be to identify predictors of achieving drug interaction score reductions after switching to a BIC/TAF/FTC-based ART regimen. Predictors for achieving drug interaction score reductions will be examined using a multivariable linear regression model. Initial models will include all a priori determined variables and all variables will be examined for multi-collinearity. Models will be fit using a backwards selection procedure. Candidate predictors will be eliminated individually by comparing the log likelihood ratio test for each model step and using the 5% significance level.

ELIGIBILITY:
Inclusion Criteria:

1. HIV diagnosis
2. 18 years of age or older
3. Receiving ART for at least 3 months
4. ART is switched to bictegravir/emtricitabine/tenofovir alafenamide between 2/7/2018 and 3/30/2019
5. Patient is receiving at least one chronic or as needed non-ART medication at the time of the switch

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults living with HIV infection and receiving antiretroviral therapy who have changed treatments to bictegravir/emtricitabine/tenofovir alafenamide
Sampling Method: Non-Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-05 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
Changes in drug interactions after switching to bictegravir/emtricitabine/tenofovir alafenamide | 1 year
  The primary endpoint is to measure the change in mean total drug interaction scores pre and post ART switch to a bictegravir/emtricitabine/tenofovir alafenamide-based regimen. The total drug interaction scores for each patient pre- and post-switch will be calculated using a drug interaction score developed for this study. The score is obtained when entering a patient's ART and concomitant medications (CM) into the University of Liverpool's HIV Drug Interaction Checker database [21]. Each ART-CM pair is given one of the following scores: "do not co-administer" is a score of 2, "potential interaction" a score of 1, and "potential weak interaction" or "no interaction" a score of 0. When no interactions are observed between a patient's ART and CMs, the total score will be 0. Higher scores occur when interactions are present. A decrease in score indicates that switching to bictegravir/emtricitabine/tenofovir alafenamide decreased the number and severity of interactions present.

SECONDARY OUTCOMES:
Predictors of achieving drug interaction score reductions after switching to bictegravir/emtricitabine/tenofovir alafenamide | 1 year
  The secondary endpoint of the study is to identify predictors of drug interaction score reductions after switching to a bictegravir/emtricitabine/tenofovir alafenamide. Predictors will be examined using multivariable linear regression. Initial models will include all a priori variables which will be examined for multi-collinearity. Models will be fit using a backwards selection procedure. Candidate predictors will be eliminated individually by comparing the log likelihood ratio test for each model step and using the 5% significance level.

CONTACTS AND LOCATIONS:
Overall Officials: Jason J Schafer, PharmD, MPH, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saag MS, Benson CA, Gandhi RT, Hoy JF, Landovitz RJ, Mugavero MJ, Sax PE, Smith DM, Thompson MA, Buchbinder SP, Del Rio C, Eron JJ Jr, Fatkenheuer G, Gunthard HF, Molina JM, Jacobsen DM, Volberding PA. Antiretroviral Drugs for Treatment and Prevention of HIV Infection in Adults: 2018 Recommendations of the International Antiviral Society-USA Panel. JAMA. 2018 Jul 24;320(4):379-396. doi: 10.1001/jama.2018.8431. PMID 30043070
- [Background] Beer L, Skarbinski J. Adherence to antiretroviral therapy among HIV-infected adults in the United States. AIDS Educ Prev. 2014 Dec;26(6):521-37. doi: 10.1521/aeap.2014.26.6.521. PMID 25490733
- [Background] Pantuzza LL, Ceccato MDGB, Silveira MR, Junqueira LMR, Reis AMM. Association between medication regimen complexity and pharmacotherapy adherence: a systematic review. Eur J Clin Pharmacol. 2017 Nov;73(11):1475-1489. doi: 10.1007/s00228-017-2315-2. Epub 2017 Aug 4. PMID 28779460
- [Background] Yager J, Faragon J, McGuey L, Hoye-Simek A, Hecox Z, Sullivan S, Neubert S, Patel N. Relationship Between Single Tablet Antiretroviral Regimen and Adherence to Antiretroviral and Non-Antiretroviral Medications Among Veterans' Affairs Patients with Human Immunodeficiency Virus. AIDS Patient Care STDS. 2017 Sep;31(9):370-376. doi: 10.1089/apc.2017.0081. Epub 2017 Aug 3. PMID 28771023
- [Background] Lennox JL, DeJesus E, Lazzarin A, Pollard RB, Madruga JV, Berger DS, Zhao J, Xu X, Williams-Diaz A, Rodgers AJ, Barnard RJ, Miller MD, DiNubile MJ, Nguyen BY, Leavitt R, Sklar P; STARTMRK investigators. Safety and efficacy of raltegravir-based versus efavirenz-based combination therapy in treatment-naive patients with HIV-1 infection: a multicentre, double-blind randomised controlled trial. Lancet. 2009 Sep 5;374(9692):796-806. doi: 10.1016/S0140-6736(09)60918-1. Epub 2009 Aug 3. PMID 19647866
- [Background] DeJesus E, Rockstroh JK, Henry K, Molina JM, Gathe J, Ramanathan S, Wei X, Yale K, Szwarcberg J, White K, Cheng AK, Kearney BP; GS-236-0103 Study Team. Co-formulated elvitegravir, cobicistat, emtricitabine, and tenofovir disoproxil fumarate versus ritonavir-boosted atazanavir plus co-formulated emtricitabine and tenofovir disoproxil fumarate for initial treatment of HIV-1 infection: a randomised, double-blind, phase 3, non-inferiority trial. Lancet. 2012 Jun 30;379(9835):2429-2438. doi: 10.1016/S0140-6736(12)60918-0. PMID 22748590
- [Background] Sax PE, DeJesus E, Mills A, Zolopa A, Cohen C, Wohl D, Gallant JE, Liu HC, Zhong L, Yale K, White K, Kearney BP, Szwarcberg J, Quirk E, Cheng AK; GS-US-236-0102 study team. Co-formulated elvitegravir, cobicistat, emtricitabine, and tenofovir versus co-formulated efavirenz, emtricitabine, and tenofovir for initial treatment of HIV-1 infection: a randomised, double-blind, phase 3 trial, analysis of results after 48 weeks. Lancet. 2012 Jun 30;379(9835):2439-2448. doi: 10.1016/S0140-6736(12)60917-9. PMID 22748591
- [Background] DeJesus E, Rockstroh JK, Lennox JL, Saag MS, Lazzarin A, Zhao J, Wan H, Rodgers AJ, Walker ML, Miller M, DiNubile MJ, Nguyen BY, Teppler H, Leavitt R, Sklar P; STARTMRK Investigators. Efficacy of raltegravir versus efavirenz when combined with tenofovir/emtricitabine in treatment-naive HIV-1-infected patients: week-192 overall and subgroup analyses from STARTMRK. HIV Clin Trials. 2012 Jul-Aug;13(4):228-32. doi: 10.1310/hct1304-228. PMID 22849964
- [Background] Raffi F, Jaeger H, Quiros-Roldan E, Albrecht H, Belonosova E, Gatell JM, Baril JG, Domingo P, Brennan C, Almond S, Min S; extended SPRING-2 Study Group. Once-daily dolutegravir versus twice-daily raltegravir in antiretroviral-naive adults with HIV-1 infection (SPRING-2 study): 96 week results from a randomised, double-blind, non-inferiority trial. Lancet Infect Dis. 2013 Nov;13(11):927-35. doi: 10.1016/S1473-3099(13)70257-3. Epub 2013 Sep 25. PMID 24074642
- [Background] Sax PE, Pozniak A, Montes ML, Koenig E, DeJesus E, Stellbrink HJ, Antinori A, Workowski K, Slim J, Reynes J, Garner W, Custodio J, White K, SenGupta D, Cheng A, Quirk E. Coformulated bictegravir, emtricitabine, and tenofovir alafenamide versus dolutegravir with emtricitabine and tenofovir alafenamide, for initial treatment of HIV-1 infection (GS-US-380-1490): a randomised, double-blind, multicentre, phase 3, non-inferiority trial. Lancet. 2017 Nov 4;390(10107):2073-2082. doi: 10.1016/S0140-6736(17)32340-1. Epub 2017 Aug 31. PMID 28867499
- [Background] Arribas JR, Pialoux G, Gathe J, Di Perri G, Reynes J, Tebas P, Nguyen T, Ebrahimi R, White K, Piontkowsky D. Simplification to coformulated elvitegravir, cobicistat, emtricitabine, and tenofovir versus continuation of ritonavir-boosted protease inhibitor with emtricitabine and tenofovir in adults with virologically suppressed HIV (STRATEGY-PI): 48 week results of a randomised, open-label, phase 3b, non-inferiority trial. Lancet Infect Dis. 2014 Jul;14(7):581-9. doi: 10.1016/S1473-3099(14)70782-0. Epub 2014 Jun 5. PMID 24908551
- [Background] Huhn GD, Tebas P, Gallant J, Wilkin T, Cheng A, Yan M, Zhong L, Callebaut C, Custodio JM, Fordyce MW, Das M, McCallister S. A Randomized, Open-Label Trial to Evaluate Switching to Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide Plus Darunavir in Treatment-Experienced HIV-1-Infected Adults. J Acquir Immune Defic Syndr. 2017 Feb 1;74(2):193-200. doi: 10.1097/QAI.0000000000001193. PMID 27753684
- [Background] Tsiang M, Jones GS, Goldsmith J, Mulato A, Hansen D, Kan E, Tsai L, Bam RA, Stepan G, Stray KM, Niedziela-Majka A, Yant SR, Yu H, Kukolj G, Cihlar T, Lazerwith SE, White KL, Jin H. Antiviral Activity of Bictegravir (GS-9883), a Novel Potent HIV-1 Integrase Strand Transfer Inhibitor with an Improved Resistance Profile. Antimicrob Agents Chemother. 2016 Nov 21;60(12):7086-7097. doi: 10.1128/AAC.01474-16. Print 2016 Dec. PMID 27645238
- [Background] McNicholl IR, Gandhi M, Hare CB, Greene M, Pierluissi E. A Pharmacist-Led Program to Evaluate and Reduce Polypharmacy and Potentially Inappropriate Prescribing in Older HIV-Positive Patients. Pharmacotherapy. 2017 Dec;37(12):1498-1506. doi: 10.1002/phar.2043. Epub 2017 Nov 30. PMID 29023938
- [Background] Gallant J, Hsue PY, Shreay S, Meyer N. Comorbidities Among US Patients With Prevalent HIV Infection-A Trend Analysis. J Infect Dis. 2017 Dec 19;216(12):1525-1533. doi: 10.1093/infdis/jix518. PMID 29253205
- [Background] Nachega JB, Mugavero MJ, Zeier M, Vitoria M, Gallant JE. Treatment simplification in HIV-infected adults as a strategy to prevent toxicity, improve adherence, quality of life and decrease healthcare costs. Patient Prefer Adherence. 2011;5:357-67. doi: 10.2147/PPA.S22771. Epub 2011 Jul 18. PMID 21845035
- [Background] Iniesta-Navalon C, Franco-Miguel JJ, Gascon-Canovas JJ, Rentero-Redondo L. Identification of potential clinically significant drug interactions in HIV-infected patients: a comprehensive therapeutic approach. HIV Med. 2015 May;16(5):273-9. doi: 10.1111/hiv.12205. Epub 2014 Dec 18. PMID 25523089
- [Background] So-Ngern A, Montakantikul P, Manosuthi W. Clinically significant drug interactions among HIV-infected patients receiving antiretroviral therapy. Southeast Asian J Trop Med Public Health. 2014 Sep;45(5):1023-31. PMID 25417503
- [Background] Miller CD, El-Kholi R, Faragon JJ, Lodise TP. Prevalence and risk factors for clinically significant drug interactions with antiretroviral therapy. Pharmacotherapy. 2007 Oct;27(10):1379-86. doi: 10.1592/phco.27.10.1379. PMID 17896893
- See also: HIV Drug Interactions. University of Liverpool. — https://www.hiv-druginteractions.org/